CLINICAL TRIAL: NCT00595842
Title: Clinical Success of Artificial Root-End Barriers With Mineral Trioxide Aggregate in Teeth With Immature Apices
Brief Title: Artificial Root-End Barriers
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: 59th Medical Wing (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kenneth Hargreaves, Chair, Dept. of Endodontics, The University of Texas Health Science Center at San Antonio
Other Study IDs: HSC20070204
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Dental Cements; Tooth Abnormalities
Keywords: Mineral trioxide aggregate
MeSH Terms: conditions — Tooth Abnormalities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group one: Subjects are drawn from a search of all patients treated with MTA between ages 5-40

SUMMARY:
This study retrospectively looks to determine the clinical success of ProRoot MTA used as an artificial apical barrier in teeth with immature apices.

DETAILED DESCRIPTION:
The normal development and maturation of a root depends on a vital, healthy pulp. If the pulp becomes necrotic in a tooth with an immature apex, endodontic treatment can be performed using an artificial barrier technique. Mineral trioxide aggregate (MTA) has become the material of choice to accomplish this procedure, however, few studies have evaluated its clinical success. The purpose of this retrospective study was to determine the clinical success of ProRoot MTA used as an artificial apical barrier. Twenty patients were included in this study. After approximately one week of Ca(OH)2 treatment, each patient had MTA placed as an apical barrier in a tooth with a single canal and open apex followed by placement of a final restoration. Patients were recalled and evaluated for clinical signs and symptoms and osseous healing. Immediate post-treatment and recall radiographs were evaluated by two endodontists calibrated for use of the Periapical Index (PAI).

ELIGIBILITY:
Inclusion Criteria:

* a tooth with a single canal and presence of an open apex by radiograph
* Ca(OH)2 treatment for at least one week prior to obturation
* use of MTA to produce an artificial apical barrier
* placement of a final restoration
* radiographs codumenting pretreatment and immedicate post-treatment conditionof the tooth
* patients ages 5-40 years old

Exclusion Criteria:

* patients younger than 5 and greater than 40 years old
* patients unable to be contacted for recall during the study
* patients with a medical condition whose health would be jeopardized by participation in the study

Ages: 5 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients between 5-40 years old who have been treated with MTA
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2007-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Holden, DMD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Health Science Center, San Antonio, Texas, United States